CLINICAL TRIAL: NCT01967147
Title: Evaluation of Clinical Outcomes Following Treatment With Systane® Balance in Dry Eye Subjects With Lipid Deficiency
Brief Title: Clinical Outcomes Following Treatment With Systane® Balance in Dry Eye Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-13-027
Record Dates: First submitted 2013-10-18; First posted 2013-10-22 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Dry Eye
Keywords: Dry eye; Lipid deficiency; Tear film break-up time
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Propylene Glycol; Ophthalmic Solutions; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Balance (Experimental): Propylene Glycol, 0.6% eye drops, 1 drop in each eye, 4 times per day, during Phase I (Day 0-35), followed by 1 drop in each eye as needed during Phase II (Day 35-90).
  Interventions: Drug: Propylene Glycol, 0.6% eye drops
- Saline (Active Comparator): Preservative-Free 0.9% Saline solution, 1 drop in each eye, 4 times per day, during Phase I (Day 0-35), followed by 1 drop in each eye as needed during Phase II (Day 35-90).
  Interventions: Drug: Preservative-free 0.9% Saline solution

INTERVENTIONS:
Drug: Propylene Glycol, 0.6% eye drops — Commercially available eye drops used during Treatment Phase
  Other Names: Systane® Balance
  Arms: Systane Balance
Drug: Preservative-free 0.9% Saline solution — Commercially available solution used as Run-in (1 drop in each eye 4 times a day for 15 days) and during Treatment Phase
  Arms: Saline

SUMMARY:
The purpose of this study is to demonstrate the superior efficacy of Systane® Balance over Preservative-Free 0.9% Saline following 35 days of QID (4 times a day) dosing in treating dry eye subjects with lipid deficiency.

DETAILED DESCRIPTION:
This study consisted of 4 visits conducted during 3 sequential phases: the Run-in Phase (which included a screening visit and run-in period), Treatment Phase I and Treatment Phase II. In Phase I, subjects were randomized to either Systane® Balance or Saline and dosed 4 times a day for 35 days. In Phase II (Day 35-90) subjects continued to dose with their assigned product on an as-needed basis.

ELIGIBILITY:
Inclusion Criteria:

* Must have all of the following in at least 1 eye at Screening:

  1. Meibomian Gland Dysfunction (MGD) grading for Expressibility ≤ 2 and Meibum Quality ≤ 2,
  2. The average of 3 measures of TFBUT ≤ 5 seconds, and
  3. Unanesthetized Schirmer I test of ≥ 3 mm.
* Must have an Ocular Surface Disease Index (OSDI) Score ≥ 18 at Visit 1 prior to randomization (ie, after 2 weeks of run-in with Preservative-Free 0.9% Saline administered 4 times a day).
* Must have best-corrected visual acuity of 55 letters or better in each eye as assessed using an early treatment diabetic retinopathy study (ETDRS) chart (letter read method).
* Physician diagnosis of dry eye at least 6 months prior to Screening visit.
* Willing and able to attend all study visits.
* Must sign a written informed consent form.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Subjects on topical ocular treatments containing benzalkonium chloride (BAK), or other products with known toxicity to the corneal surface, within 30 days of Screening.
* Subjects who have started, stopped, or changed a lid hygiene regimen within 30 days of Screening.
* Use of any artificial tears/lubricants/gels/rewetting drops within 4 hours of Screening.
* Women of childbearing potential are excluded from participating in this study if they met any of the following conditions:

  * Currently pregnant, or
  * Test positive for pregnancy at Screening visit, or
  * Currently breast feeding, or
  * Are not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.
* Hypersensitivity to the use of any of the study products or allergy to any ingredient in the study products.
* Has an active ocular allergy.
* Any ocular abnormalities that could adversely affect the safety or efficacy outcome, including eyelid anomalies, corneal disorders, history of herpes simplex, etc.
* Subjects taking any systemic medication known to cause dry eye unless they have been on stable therapy/dosage for at least 30 days prior to Screening and will remain on a stable dosage for the duration of the study.
* History of any ocular or intraocular surgery (including periocular Botox injections), eyelid surgery, keratorefractive procedure, corneal transplant and its variants, or serious ocular trauma within 1 year of Screening.
* Active ocular infection (bacterial, viral or fungal), active inflammation not associated with dry eye such as uveitis, iritis, active blepharitis, active allergic conjunctivitis, etc.
* Subjects with punctal plug insertion or diathermy procedure initiated within 30 days of Screening.
* Any significant illnesses that could be expected to interfere with the study parameters.
* Subjects with active oculodermal rosacea with meibomian gland dysfunction.
* Participation in an investigational drug or device trial within 30 days of Screening.
* Contact lens use within 30 days prior to Screening, or unwilling to avoid contact lens use during the course of the study.
* Unwilling to avoid the use of additional artificial tears/lubricants/gels/rewetting drops (other than the assigned study medication) throughout the course of the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Clinical Manager, GCRA, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 14 study centers located in France, 4 study centers located in Germany, 3 study centers located in Spain, 3 study centers located in the Netherlands, 4 study centers located in the UK, 4 study centers located in Italy, and 3 study centers located in Poland.
Pre-assignment Details: Of the 279 subjects enrolled, 40 were exited as screen failures prior to randomization. An additional 25 were discontinued prior to randomization, following the outcome of the interim analysis. This reporting group includes all randomized subjects (214).
Groups:
- Systane Balance: Propylene Glycol, 1 drop in each eye, 4 times per day, during Phase I, followed by 1 drop in each eye as needed during Phase II
- Saline: Saline solution, 1 drop in each eye, 4 times/day, during Phase I, followed by 1 drop in each eye as needed during Phase II
Period: Overall Study
Arm/Group | Systane Balance | Saline
Started | 112 | 102
Completed | 99 | 82
Not Completed | 13 | 20
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 1 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Non-compliance with Study Drug | 0 | 3
Not completed — Other | 4 | 5

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Balance | Saline | Total
Number analyzed (Participants) | 112 | 102 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (15.5) | 58.4 (14.0) | 59.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 72 | 163
  Male | 21 | 30 | 51
Tear Film Break-up Time (TFBUT) [Mean (Standard Deviation); unit: seconds] | 3.73 (1.37) | 3.71 (1.59) | 3.72 (1.48)
Total Ocular Surface Staining (TOSS) Score [Mean (Standard Deviation); unit: units on a scale] — The TOSS score (a cumulative cornea and conjunctival staining score) was assessed by the investigator using ophthalmic dye and a biomicroscope. Three areas of the ocular surface were graded for dryness on a 0-5 scale (0=Absent, 5=Severe), with a resultant overall score of 0-15.
  units on a scale | 3.45 (2.14) | 3.35 (2.38) | 3.40 (2.25)
Ocular surface disease index (OSDI) [Mean (Standard Deviation); unit: units on a scale] — The OSDI is a 12-item quality of life questionnaire designed to assess ocular surface symptoms, their severity, and their impact on the subject's ability to function. Each item was scored by the subject on a 0-4 Likert-type scale (0=None, 4=All of the Time), with a resultant overall score of 0-100 (0=no disability, 100=complete disability).
  units on a scale | 40.24 (17.48) | 38.27 (17.39) | 39.30 (17.42)
Impact of Dry Eye on Everyday Life (IDEEL) Treatment Effectiveness Score [Mean (Standard Deviation); unit: units on a scale] — The IDEEL is a 10-item questionnaire designed to assess the subject's general satisfaction with treatment use. The subject responded to treatment effectiveness questions (Questions 2-5) using a 0-4 Likert-type scale, where 0=None of the time and 4=All of the time. The IDEEL treatment effectiveness score was calculated as the sum of the responses from Questions 2-5 divided by the number of questions (2-5) answered, multiplied by 25, for a resultant overall score of 0-100.
  units on a scale | 44.63 (27.32) | 46.15 (27.86) | 45.35 (27.52)
IDEEL Treatment Inconvenience [Mean (Standard Deviation); unit: units on a scale] — The IDEEL is a 10-item questionnaire designed to assess the subject's general satisfaction with treatment use. The subject responded to treatment inconvenience questions (Questions 6, 8-10) using a 0-4 Likert-type scale, where 0=All of the time and 4=None of the time. The IDEEL treatment inconvenience score was calculated as the sum of the responses from Questions 6, 8-10 divided by the number of questions (6, 8-10) answered, multiplied by 25, for a resultant overall score of 0-100.
  units on a scale | 76.61 (22.08) | 74.48 (24.85) | 75.60 (23.40)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in TFBUT at Day 35
Description: TFBUT (the time required for dry spots to appear on the corneal surface after blinking) was assessed by the investigator using ophthalmic dye and a biomicroscope and measured in seconds. Subjects were dosed in the office 1 hour ±10 minutes prior to TFBUT assessment. A shorter TFBUT indicates a higher likelihood of dry eye symptoms. A positive change indicates an improvement in TFBUT. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 35
Population: This analysis population includes all randomized subjects.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Systane Balance | Saline
Number analyzed (Participants) | 112 | 102
seconds | 1.5 (0.2) | 0.5 (0.2)

2. Secondary Outcome: Change From Baseline in TOSS Score at Day 35
Description: The TOSS score (a cumulative cornea and conjunctival staining score) was assessed by the investigator using ophthalmic dye and a biomicroscope. Three areas of the ocular surface were graded for dryness on a 0-5 scale (0=Absent, 5=Severe), with a resultant overall score of 0-15. A negative change indicates an improvement in dry eye-related staining. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 35
Population: This analysis population includes all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Systane Balance | Saline
Number analyzed (Participants) | 112 | 102
units on a scale | -0.81 (0.14) | -0.64 (0.15)

3. Secondary Outcome: Change From Baseline in OSDI Score at Day 35
Description: The OSDI is a 12-item quality of life questionnaire designed to assess ocular surface symptoms, their severity, and their impact on the subject's ability to function. Each item was scored by the subject on a 0-4 Likert-type scale (0=None, 4=All of the Time), with a resultant overall score of 0-100 (0=no disability, 100=complete disability). A negative change number represents a perceived improvement in ocular health.
Time Frame: Baseline (Day 0), Day 35
Population: This analysis population includes all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Systane Balance | Saline
Number analyzed (Participants) | 112 | 102
units on a scale | -13.7 (1.44) | -8.38 (1.56)

4. Secondary Outcome: Change From Baseline in IDEEL Treatment Effectiveness Score at Day 35
Description: The IDEEL is a 10-item questionnaire designed to assess the subject's general satisfaction with treatment use. The subject responded to treatment effectiveness questions (Questions 2-5) using a 0-4 Likert-type scale, where 0=None of the time and 4=All of the time. The IDEEL treatment effectiveness score was calculated as the sum of the responses from Questions 2-5 divided by the number of questions (2-5) answered, multiplied by 25, for a resultant overall score of 0-100. A positive change number represents perceived improvement.
Time Frame: Baseline (Day 0), Day 35
Population: This analysis population includes all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Systane Balance | Saline
Number analyzed (Participants) | 112 | 102
units on a scale | 21.51 (2.43) | 5.50 (2.65)

5. Secondary Outcome: Change From Baseline in IDEEL Treatment Inconvenience Score at Day 35
Description: The IDEEL is a 10-item questionnaire designed to assess the subject's general satisfaction with treatment use. The subject responded to treatment inconvenience questions (Questions 6, 8-10) using a 0-4 Likert-type scale, where 0=All of the time and 4=None of the time. The IDEEL treatment inconvenience score was calculated as the sum of the responses from Questions 6, 8-10 divided by the number of questions (6, 8-10) answered, multiplied by 25, for a resultant overall score of 0-100. A positive change number represents perceived improvement.
Time Frame: Baseline (Day 0), Day 35
Population: This analysis population includes all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Systane Balance | Saline
Number analyzed (Participants) | 112 | 102
units on a scale | 1.30 (1.56) | 0.77 (1.70)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 90 days). AEs were reported as pretreatment and treatment-emergent. Ocular adverse events are presented for both study eye and non-study eye.
Description: An AE was defined as any untoward medical occurrence, unintended injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the medical device/product. AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the Investigator, as outlined in the protocol.
Groups:
- Pretreatment: All subjects prior to exposure to investigational product
- Systane Balance: All subjects exposed to Systane® Balance
- Saline: All subjects exposed to Saline
Arm/Group | Pretreatment | Systane Balance | Saline
Serious Adverse Events (participants affected / at risk) | 0/279 | 2/110 | 2/100
Other Adverse Events (participants affected / at risk) | 0/279 | 6/110 | 1/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=279) | Systane Balance (N=110) | Saline (N=100)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal cyst excision (Surgical and medical procedures) | 0 | 0 | 1
Laryngeal operation (Surgical and medical procedures) | 0 | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=279) | Systane Balance (N=110) | Saline (N=100)
Eye irritation (Eye disorders) | 0 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.